CLINICAL TRIAL: NCT07071415
Title: Breast Cancer Screening Decision Aid
Brief Title: Overdiagnosis and Breast Cancer Screening Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2000040131; K08CA248725 (NIH)
Record Dates: First submitted 2025-06-21; First posted 2025-07-17 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Mammography Screening; Geriatrics; Decision Aid
Keywords: breast cancer screening; health-related beliefs; overdiagnosis; mammography; older women

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low risk of overdiagnosis (Experimental): Participants in this arm will be shown a decision aid in which risk of overdiagnosis is low.
  Interventions: Behavioral: Breast cancer screening decision aid -- low risk
- Moderate risk of overdiagnosis (Experimental): Participants in this arm will be shown a decision aid in which risk of overdiagnosis is moderate.
  Interventions: Behavioral: Breast cancer decision aid -- moderate risk
- High risk of overdiagnosis (Experimental): Participants in this arm will be shown a decision aid in which risk of overdiagnosis is high.
  Interventions: Behavioral: Breast cancer screening decision aid -- high risk
- Control (Active Comparator): Participants in this arm will be shown a video about breast cancer screening that is identical in all ways but contains no information about overdiagnosis.
  Interventions: Other: Control condition

INTERVENTIONS:
Behavioral: Breast cancer screening decision aid -- low risk — Participants in this study will view a video-based decision aid that describes the risks and benefits of breast cancer screening for older women. Participants assigned to the low risk of overdiagnosis arm will view a version of the decision aid the describes a low risk of overdiagnosis.
  Arms: Low risk of overdiagnosis
Behavioral: Breast cancer decision aid -- moderate risk — Participants in this study will view a video-based decision aid that describes the risks and benefits of breast cancer screening for older women. Participants assigned to the moderate risk of overdiagnosis arm will view a version of the decision aid the describes a moderate risk of overdiagnosis.
  Arms: Moderate risk of overdiagnosis
Behavioral: Breast cancer screening decision aid -- high risk — Participants in this study will view a video-based decision aid that describes the risks and benefits of breast cancer screening for older women. Participants assigned to the high risk of overdiagnosis arm will view a version of the decision aid the describes a high risk of overdiagnosis.
  Arms: High risk of overdiagnosis
Other: Control condition — Participants in this study will view a video-based decision aid that describes the risks and benefits of breast cancer screening for older women. Participants assigned to the control arm will view a version of the decision aid that does not contain any information about overdiagnosis.
  Arms: Control

SUMMARY:
This is a survey-based study using an online panel. The goal of the study is to understand whether information about overdiagnosis influences breast cancer screening intention among older women. Participants are first asked a series of questions about breast cancer screening including their intention to continue screening, knowledge of screening, and beliefs about screening. They are then shown one of three videos about breast cancer screening that contain information about overdiagnosis or a fourth control video that is identical but contains no information about overdiagnosis. Participants are then again asked about screening intention, along with knowledge of screening, overdiagnosis, and questions around trust.

ELIGIBILITY:
Inclusion Criteria:

* 70 and older
* Able to participate in an English-language web-based survey

Exclusion Criteria:

* Prior history of breast cancer or ductal carcinoma in situ

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 311 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Participants intention to screen | Day 1
  Intention to screen, measured on a 15 point scale. Total score range 1-15, lower score means less likely to screen.

SECONDARY OUTCOMES:
Knowledge of breast cancer screening | Day 1
  Knowledge of screening will be quantified as the proportion of correct answers out of a total possible 7 questions in the pre test and 11 questions in the post test.
Understanding of overdiagnosis | Day 1
  Understanding of overdiagnosis will be quantified as proportion of correct responses out of 3 questions about overdiagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Richman, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Supporting information is available immediately from investigators. Individual patient data will be available beginning one year after data collection.
Access Criteria: Available to qualified researchers upon request.